CLINICAL TRIAL: NCT04885816
Title: Drug-Eluting Balloon Versus Drug-eluting Stent On de Novo coRonary Artery Disease in Patients With High Bleeding Risk
Brief Title: Drug-eluting Balloon Versus Drug-eluting Stent for High Bleeding Risk Angioplasty
Acronym: DEBORA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Daniel Fernando Zazueta Salido, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INCAR-DG-DACEP-020-2021; 21-1223 (Other: INCar Protocol Number)
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: High Bleeding Risk; Coronary Artery Disease (CAD); Percutaneous Coronary Intervention (PCI)
Keywords: Drug Eluting Balloon (DEB); Drug Eluting Stent (DES); High bleeding risk (HBR); High hemorrhagic risk; Dual anti-platelet therapy (DAPT)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, non-inferiority clinical trial enrolling high bleeding risk patients and coronary artery disease to be treated by percutaneous coronary intervention at the National Institute of Cardiology "Ignacio Chávez" in México. Included patients will have follow-up at the outpatient clinic through 1 year, until death or study exit, whichever comes first.
Who Masked: Participant
Masking Description: Randomized treatment will not be revealed to patient at any time during procedure or afterwards until follow-up is done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Eluting Balloon (DEB) (Experimental): High Bleeding Risk patients treated with 2.5 - 4.0 mm drug-eluting balloons (DEB). Bailout stenting is permitted in case of a flow-limiting dissection or significant recoil (>30% in main branch and >50% side-branch), includes both stable coronary artery disease (SCAD) and acute coronary syndromes (ACS) patients undergoing elective Percutaneous Coronary Intervention (PCI).
  Interventions: Device: Drug Eluting Balloon (DEB)
- Drug Eluting Stents (DES) (Active Comparator): High Bleeding Risk patients treated with 2.5 - 4.0 mm drug-eluting stents (DES). Includes both stable CAD and ACS patients undergoing elective PCI.
  Interventions: Device: Drug Eluting Stents (DES)

INTERVENTIONS:
Device: Drug Eluting Balloon (DEB) — Size (diameter and length) will be chosen at operator's discretion aid by simple angiography, quantitative coronary analysis (QCA), or intravascular image; so that the lesion previously prepared and 2 mm at each end are covered by DEB, and the diameter and pressure used aims a balloon to artery ratio of 1. In case of significant recoil (more than 30% for main vessels and 50% for side vessels), coronary perforation or flow limiting dissection, provisional stent will be implanted with a stent to artery ratio of 1.1 with stent post-dilatation when indicated. Device will be used in accordance with the CE mark instructions.
  DAPT will be given for a month with aspirin and a P2Y12 inhibitor (clopidogrel will be favored). Single anti-platelet therapy (SAPT) with aspirin will be continued thereafter.
  Other Names: MagicTouch, Sirolimus coated balloon catheter, diameters 2.5 - 4.0 mm (Concept Medicals, Surat, India)
  Arms: Drug Eluting Balloon (DEB)
Device: Drug Eluting Stents (DES) — Size (diameter and length) will be chosen at operator's discretion aid by simple angiography, quantitative coronary analysis (QCA), or intravascular image; so that the lesion previously prepared and 2 mm at each end are covered by DES with an stent to artery ratio of 1.1. Post-dilatation will be performed when indicated. Devices will be used in accordance with the CE mark instructions.
  DAPT will be indicated according to actual international guidelines.
  Other Names: Orsiro, Sirolimus eluting stent, diameters 2.5 - 4.0 mm (Biotronik AG, Bülach, Switzerland); Resolute Onyx, Zotarolimus eluting stent, diameters 2.5 - 4.0 mm (Medtronic, Santa Rosa, CA, USA); Xiencie Sierra, Everolimus eluting stent, diameters 2.5 - 4.0 mm (Abbott Vascular, Santa Clara, CA, USA); Synergy, Everolimus eluting stent, diameters 2.5 - 4.0 mm (Boston Scientific, Natick, MA, USA)
  Arms: Drug Eluting Stents (DES)

SUMMARY:
Randomized, single-blind, single-center, non-inferiority clinical trial to compare target lesion failure (TLF) at 12 months in high bleeding risk patients undergoing elective coronary percutaneous intervention comparing limus-eluting balloon vs. limus-eluting stents.

DETAILED DESCRIPTION:
Drug Eluting Stents (DES) are the devices of choice for coronary angioplasty, including in patients with high-bleeding risk.

Different studies have been done to determine which strategy improves bleeding outcomes without risking the benefit of stenting. Different Double Anti-Platelet Therapy (DAPT) durations in different devices have shown that it is safe to reduce DAPT, with an increase in ischemic events but a better net clinical outcome.

Safety and efficacy of Drug Eluting Balloons (DEB) were proved when it was compared with Bare Metal Stents (BMS) in de-novo coronary lesions by presenting no events of target vessel closure after treatment.

Our hypothesis is that treating this group of high-bleeding risk patients with DEB will be no-inferior in terms of target vessel failure at 12 months when compared with DES for treatment of de-novo coronary lesions in high bleeding risk population, reducing incidence of significant bleeding events with DAPT reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older with an ischemic de-novo lesion(s) in a 2.5 - 4.0 mm reference diameter coronary artery suitable for elective percutaneous coronary intervention, in context of acute coronary syndrome or chronic coronary syndrome with evidence of ischemia by non-invasive study or pressure guidewire that can be treated by DEB or DES, and has at least 1 major or 2 minor Academic Research Consortium High Bleeding Risk criteria:
* Major criteria:

  1. Anticipated use of long-term oral anticoagulation
  2. Severe or end-stage CKD (eGFR <30 mL/min)
  3. Hemoglobin < 11 g/dL
  4. Spontaneous bleeding requiring hospitalization or transfusion in the last 6 months, or any time, if recurrent.
  5. Moderate or severe baseline thrombocytopenia (<100,000/uL)
  6. Chronic bleeding diathesis
  7. Liver cirrhosis with portal hypertension
  8. Active malignancy (excluding nonmelanoma skin cancer) within the past 12 months
  9. Previous spontaneous intracranial hemorrhage
  10. Previous traumatic intracranial hemorrhage within the past 12 months
  11. Presence of Brain arteriovenous malformation (AVM)
  12. Moderate or severe ischemic stroke (NIHSS score equal or more than 5) within the past 6 months
  13. Non deferrable major surgery while on DAPT
  14. Recent major surgery or major trauma within 30 days before PCI
* Minor Criteria:

  1. Age 75 years old and older
  2. Moderate Chronic Kidney Disease (CKD) (eGFR 30-59 mL/min)
  3. Hemoglobin 11 - 12.9 g/dL in men and 11 - 11.9 g/dL in women
  4. Spontaneous bleeding requiring hospitalization or transfusion within the past 12 months, not meeting major criterion
  5. Long term use of NSAIDs or steroids
  6. Any ischemic stroke at any time not meeting major criterion

Exclusion Criteria:

* STEMI undergoing primary PCI
* Any ACS undergoing urgent PCI
* Cardiogenic shock or resuscitation with uncertain neurological status at arrival to PCI
* Unprotected left main lesion
* Life expectancy < 12 months
* Reference vessel diameter < 2.5 mm or > 4.0 mm
* Bifurcation lesion requiring 2-stent technique
* Chronic total occlusion
* In-stent restenosis
* Dissection affecting the flow (TIMI<3) or significant recoil (>30% in main branch, >50% in side branch) after predilatation
* Inability to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target lesion revascularization

SECONDARY OUTCOMES:
Cardiovascular death | 12 months
  Rate of death resulting from cardiovascular causes in each group:
  Death caused by acute MI Death caused by sudden cardiac, including unwitnessed, death Death resulting from heart failure Death caused by stroke Death caused by cardiovascular procedures Death resulting from cardiovascular hemorrhage Death resulting from other cardiovascular cause Any MI not clearly attributable to a non-target vessel will be considered as target-vessel MI.
  Percutaneous coronary intervention (PCI) related MI is termed type 4a MI.
Myocardial Infarction related to the treated vessel | 12 months
  Rate of myocardial infarction related to the treated vessel (according to the 4th international definition of myocardial infarction) in each group: detection of an increase or decrease in cardiac troponin values with at least 1 of the values above the upper reference limit of the 99th percentile and at least 1 of the following conditions :
  Symptoms of acute myocardial ischemia. New ischemic changes in the electrocardiogram. Appearance of pathological Q waves. Imaging evidence of loss of viable myocardium or new regional abnormalities in myocardial wall mobility following a pattern compatible with ischemic etiology.
  Identification of a coronary thrombus by angiography with intracoronary imaging or by autopsy Any MI that cannot be clearly attributed to a vessel other than the revascularized one will be considered as MI related to the treated vessel.
Target Lesion Revascularization | 12 months
  Rate of repeated percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Target Vessel Failure (TVF) | 12 months
  Rate of TVF in each group (composed of cardiovascular death, myocardial infarction related to the treated vessel or ischemia driven target vessel revascularization)
Target Vessel Revascularization | 12 months
  Rate of repeated percutaneous intervention or surgical bypass of any segment of the target vessel in each group.
Non-cardiovascular death | 12 months
  Rate of any death that is not thought to be the result of a cardiovascular cause in each group:
  1. Death resulting from malignancy
  2. Death resulting from pulmonary causes
  3. Death caused by infection (includes sepsis)
  4. Death resulting from gastrointestinal causes
  5. Death resulting from accident/trauma
  6. Death caused by other noncardiovascular organ failure
  7. Death resulting from other noncardiovascular cause
Major Bleeding | 12 months
  Incidence of bleeding complications according to The Bleeding Academic Research Consortium 2 (BARC-2) scale: 3 or greater
Technical success | Periprocedural
  Rate of restoration of antegrade Thrombolysis In Myocardial Infarction (TIMI) flow 2 or 3 and a <30% residual stenosis.
Subgroup analysis of target lesion failure | 12 months
  Rate of TLF in treatment of bifurcations vs no bifurcation, by vessel size, in diabetes, by clinical Presentation (acute or chronic).
Subgroup analysis of major bleeding events | 12 months
  Rate of BARC 3-5 bleeding events in patients with anticoagulation vs no anticoagulation, by DAPT duration, by inclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid-Lidt, MD, Study Director — Instituto Nacional de Cardiología "Ignacio Chávez"
Locations (1):
- Instituto Nacional de Cardiologia "Ignacio Chávez", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual patient data will not be shared with other researchers.

REFERENCES:
- [Result] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Result] Kandzari DE, Kirtane AJ, Windecker S, Latib A, Kedhi E, Mehran R, Price MJ, Abizaid A, Simon DI, Worthley SG, Zaman A, Choi JW, Caputo R, Kanitkar M, McLaurin B, Potluri S, Smith T, Spriggs D, Tolleson T, Nazif T, Parke M, Lee LC, Lung TH, Stone GW; Onyx ONE US/Japan Investigators. One-Month Dual Antiplatelet Therapy Following Percutaneous Coronary Intervention With Zotarolimus-Eluting Stents in High-Bleeding-Risk Patients. Circ Cardiovasc Interv. 2020 Nov;13(11):e009565. doi: 10.1161/CIRCINTERVENTIONS.120.009565. Epub 2020 Nov 10. PMID 33167705
- [Result] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Result] Alfonso F, Scheller B. State of the art: balloon catheter technologies - drug-coated balloon. EuroIntervention. 2017 Aug 25;13(6):680-695. doi: 10.4244/EIJ-D-17-00494. PMID 28844030
- [Result] Varenne O, Cook S, Sideris G, Kedev S, Cuisset T, Carrie D, Hovasse T, Garot P, El Mahmoud R, Spaulding C, Helft G, Diaz Fernandez JF, Brugaletta S, Pinar-Bermudez E, Mauri Ferre J, Commeau P, Teiger E, Bogaerts K, Sabate M, Morice MC, Sinnaeve PR; SENIOR investigators. Drug-eluting stents in elderly patients with coronary artery disease (SENIOR): a randomised single-blind trial. Lancet. 2018 Jan 6;391(10115):41-50. doi: 10.1016/S0140-6736(17)32713-7. Epub 2017 Nov 1. PMID 29102362
- [Result] Urban P, Mehran R, Colleran R, Angiolillo DJ, Byrne RA, Capodanno D, Cuisset T, Cutlip D, Eerdmans P, Eikelboom J, Farb A, Gibson CM, Gregson J, Haude M, James SK, Kim HS, Kimura T, Konishi A, Laschinger J, Leon MB, Magee PFA, Mitsutake Y, Mylotte D, Pocock S, Price MJ, Rao SV, Spitzer E, Stockbridge N, Valgimigli M, Varenne O, Windhoevel U, Yeh RW, Krucoff MW, Morice MC. Defining High Bleeding Risk in Patients Undergoing Percutaneous Coronary Intervention. Circulation. 2019 Jul 16;140(3):240-261. doi: 10.1161/CIRCULATIONAHA.119.040167. Epub 2019 May 22. PMID 31116032
- [Result] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Result] Zocca P, Kok MM, van der Heijden LC, Danse PW, Schotborgh CE, Scholte M, Hartmann M, Linssen GCM, Doggen CJM, von Birgelen C. High Bleeding Risk Patients Treated with Very Thin-Strut Biodegradable Polymer or Thin-Strut Durable Polymer Drug-Eluting Stents in the BIO-RESORT Trial. Cardiovasc Drugs Ther. 2018 Dec;32(6):567-576. doi: 10.1007/s10557-018-6823-9. PMID 30143879